CLINICAL TRIAL: NCT05152641
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study Investigating the Efficacy and Safety of BGE-117 in Moderately to Severely Anemic Older Individuals After Major Hip Surgery
Brief Title: Study to Evaluate Efficacy and Safety of BGE-117 in Moderately to Severely Anemic Older Individuals After Major Hip Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The program priority for execution of this clinical trial changed prior to enrollment of the first patient. The study was not withdrawn due to any safety concerns.
Sponsor: BioAge Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGE-117-203
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Acute Posthemorrhagic Anemia
Keywords: Anemia; BGE-117; Hip; Surgery; Postoperative; BioAge
MeSH Terms: conditions — Anemia | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- BGE-117 4mg (Experimental): BGE-117 4mg, Capsules, Oral-administered Once Per Day up to 12 weeks Ferrous sulfate 325mg, Tablets, Oral-administered 3 Times Per Week up to 12 weeks
  Interventions: Drug: BGE-117, 4mg; Dietary Supplement: Ferrous Sulfate
- BGE-117 8mg (Experimental): BGE-117 8mg, Capsules, Oral-administered Once Per Day up to 12 weeks Ferrous sulfate 325mg, Tablets, Oral-administered 3 Times Per Week up to 12 weeks
  Interventions: Drug: BGE-117, 4mg; Dietary Supplement: Ferrous Sulfate
- BGE-117 16mg (Experimental): BGE-117 16mg, Capsules, Oral-administered Once Per Day up to 12 weeks Ferrous sulfate 325mg, Tablets, Oral-administered 3 Times Per Week up to 12 weeks
  Interventions: Drug: BGE-117, 4mg; Dietary Supplement: Ferrous Sulfate; Drug: BGE-117, 12mg
- Placebo (Placebo Comparator): Matching Placebo Capsules, Oral-administered Once Per Day up to 12 weeks Ferrous sulfate 325mg, Tablets, Oral-administered 3 Times Per Week up to 12 weeks
  Interventions: Dietary Supplement: Ferrous Sulfate; Other: Matching Placebo

INTERVENTIONS:
Drug: BGE-117, 4mg — BGE-117, 4mg Capsules
  Arms: BGE-117 16mg; BGE-117 4mg; BGE-117 8mg
Dietary Supplement: Ferrous Sulfate — Ferrous Sulfate, 325mg Tablets
Other: Matching Placebo — Matching Placebo to BGE-117 Capsules
  Arms: Placebo
Drug: BGE-117, 12mg — BGE-117, 12mg Capsules
  Arms: BGE-117 16mg

SUMMARY:
The purpose of this study is to explore the safety and tolerability of BGE-117 and gain information on the effectiveness of different doses when given to patients 65 years or older with moderate to severe anemia following major hip surgery. BGE-117 is given once daily in a capsule by mouth for up to 12 weeks. Patients are also given oral iron supplements. Anemia following surgery has been associated with decreases in patient functioning. This study will measure improvement of anemia, as well as various patient functioning.

DETAILED DESCRIPTION:
BGE-117 is being investigated to determine whether it is an effective treatment for moderate to severe anemia in older individuals (65 years of age or older) after major hip surgery. Currently, there are limited treatment options for postoperative anemia, in this patient population, available in the USA, Australia, or New Zealand. The increased risk of morbidity, mortality, and poor quality of life in the population of older individuals with postoperative anemia highlights the unmet medical need for a therapeutic agent that can alleviate physical and functional deficits in these patients. Study BGE-117-203 will be the first clinical study conducted in older patients with postoperative anemia. The study will collect important safety, efficacy, and dosing information across this population of patients to provide key data for designing further clinical studies in the development programs for BGE-117.

The study will enroll 2 populations of patients requiring hip surgery:

* older individuals who are scheduled for elective unilateral or bilateral hip surgery (total or partial hip replacement or revision of a previous replacement)
* older individuals with an acute hip fracture requiring surgical repair or replacement (usually performed within 48 hours after the fracture event)

These individuals must also meet the inclusion criterion for a hemoglobin level of ≤ 10 g/dL and ≥ 7.0 g/dL from postoperative Day 1 to postoperative Day 7.

The total planned enrollment for the study is approximately 192 subjects. The first 96 subjects who are enrolled will be randomized in a 1:2:1 ratio to 1 of 3 treatment groups:

* BGE-117 8 mg PO once daily with oral iron supplement 3 times per week (n = 24)
* BGE-117 4 mg PO once daily with oral iron supplement 3 times per week (n = 48)
* Matching placebo once daily with oral iron supplement 3 times per week (n = 24)

A Safety Review Meeting will be conducted when approximately 48 subjects have completed 4 weeks of treatment. Enrollment will remain ongoing for up to 96 subjects pending the Safety Review Meeting. If no safety concerns are identified that would preclude the inclusion of additional subjects, the subsequent 96 subjects who would be dosed up to 16 mg will be allowed to proceed without interruption. Additional safety reviews will be completed after 96 subjects and 144 subjects have completed 4 weeks of treatment.

The subsequent 96 subjects enrolled will be randomized in a 1:2:1 ratio to 1 of 3 treatment groups:

* BGE-117 8 mg PO once daily with oral iron supplement 3 times per week (n = 24)
* BGE-117 16 mg PO once daily with oral iron supplement 3 times per week (n = 48)
* Matching placebo once daily with oral iron supplement 3 times per week (n = 24)

At study completion, the goal is to have approximately 48 subjects in each of the 4 treatment groups (placebo, BGE-117 4 mg, BGE-117 8 mg, and BGE-117 16 mg) with each treatment group having a similar number of subjects with acute hip fracture or elective hip surgery.

The Treatment Period is 12 weeks, and all enrolled subjects will be followed for a total of 6 months after surgery (14 weeks after cessation of IP) to monitor hemoglobin progression and functional outcome as well as to continue to monitor for any potential AEs.

There will be no dose increases, however, dose decreases will be allowed if the rate of increase in hemoglobin exceeds the protocol defined limits. The goal is to maintain an approximate rate of hemoglobin increase of ≤ 1.5 g/dL every 2 weeks, and a maximum hemoglobin level of 12.0 g/dL. Dosing will be considered completed and no additional IP will be administered after the maximum hemoglobin value is confirmed.

Subjects will be randomized within 24 hours of meeting the hemoglobin entry criteria. The baseline hemoglobin value for the primary endpoint analysis will be the last (most recent) hemoglobin level obtained via central laboratory before administration of the first dose of blinded IP on Day 1. Treatment will start as soon as the subject has been randomized and is able to take oral medications. Subjects enrolled in the study will continue once daily treatment for a total of 12 weeks. Supplemental iron, provided by the Sponsor, will be administered orally as ferrous sulfate 325 mg 3 times per week (e.g., every Monday, Wednesday, and Friday).

Subjects may be discharged from the hospital as soon as it is medically appropriate, but they will continue to be seen at the study site at the following visits: Visit 2 (Day 1), Visit 4 (Day 15), Visit 8 (Day 43), and Visit 14 (Day 85). Home visits (including visits to rehabilitation facilities, assisted living facilities, and nursing home facilities) will be conducted at Visits 3, 5, 6, 7, 9, 10, 11, 12, and 13 to assess vital signs and collect a central blood sample for CBC and reticulocytes. There will be a home study visit approximately 14 days after administration of the last dose of IP (Visit 15). Additional home visits will be completed approximately 4 months after surgery on Day 127 (Visit 16), and approximately 5 months after surgery on Day 155 (Visit 17). A final Follow up Visit at the study site will be completed approximately 6 months after surgery on Day 183 (Visit 18).

All enrolled subjects must be able to personally give informed consent. Consent by guardian or proxy will not be permitted. Screening will include a full physical examination and baseline laboratory evaluation. Consent and screening procedures may be done preoperatively or postoperatively based on type of surgery. If a subject consents and meets eligibility criteria preoperatively, they must also meet eligibility criteria postoperatively to remain eligible for enrollment.

If a subject does not consent preoperatively (e.g., hip fracture), they can consent postoperatively. If enrolled, subjects will receive their first dose of IP at the study site. They will be instructed to take IP orally once daily, approximately 1 hour before breakfast for up to 83 additional days. Study medication will be administered in addition to oral iron supplements and standard of care as deemed appropriate by the subject's treating physicians. Oral iron in the form of ferrous sulfate 325 mg (supplied by the Sponsor) will be administered 3 times per week after an overnight fast at the same time-of-day as IP. Subjects will be monitored throughout the study for AEs and all relevant efficacy outcomes. Blood samples will be obtained periodically for safety laboratory tests, biomarkers of BGE 117 activity, inflammation, lipid, and iron status, and plasma pharmacokinetics (PK). Subjects will be followed until 6 months after their surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Alert and able to voluntarily provide written, signed, and dated informed consent
2. ≥ 65 years of age at the time of completing informed consent
3. Major hip surgery, that has occurred within the previous 7 days or is scheduled to occur within the next 7 days, defined as:

   * Unilateral or bilateral total or partial hip arthroplasty or revision OR
   * Hip fracture repair surgery scheduled or performed within 48 hours after hospital admission (either fracture repair or total or partial hip replacement)
4. Postoperative anemia defined as a hemoglobin level ≤ 10.0 g/dL and ≥ 7.0 g/dL from postoperative Day 1 to postoperative Day 7
5. For hip fracture subjects only: score between 1 and 5 on the Clinical Frailty Scale (CFS) at baseline before fracture
6. Estimated glomerular filtration rate (eGFR) of ≥ 60 mL/min/m2 as measured by the Modification of Diet in Renal Disease (MDRD) method
7. Current or planned perioperative use of mechanical or chemical antithrombotic prophylaxis in accordance with local standard of care

Exclusion Criteria:

1. Any current unstable medical condition that the investigator considers would put the subject at unacceptable risk, affect study compliance, or prevent the understanding of the study's objectives or investigational procedures or possible consequences; for example, increased risk of falls that is judged to be clinically significant, clinically significant autonomic dysfunction, active infections requiring antimicrobial treatment
2. History of thromboembolic disease in the previous 6 months
3. Other medically significant injuries (e.g., head injuries, internal bleeding, or other as judged by the study investigator) that occur concurrently with hip fractures that complicate endpoint assessments, subject safety, and/or study conduct
4. History of seizures within the previous 2 years
5. History of coagulation disorder (e.g., Factor V Leiden, idiopathic thrombocytopenic purpura) or use of concomitant medications that increase the risk of thromboembolic events (TEEs) as judged by the study investigator
6. Class III or IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system
7. QTcF > 500 msec or QTcF > 530 msec in subjects with bundle branch block. A triplicate electrocardiogram (ECG) should be performed if the initial ECG indicates prolonged QTc interval using the automated or manually calculated QTcF value.
8. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels ≥ 3 × the upper limit of normal (ULN) (Historical standard-of-care laboratory results may be used to confirm eligibility if collected within 14 days before informed consent)
9. Bilirubin level > 1.5 × ULN (isolated bilirubin level > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35%) (Historical standard of care laboratory results may be used to confirm eligibility if collected within 14 days before informed consent)
10. Recent or planned administration of an erythropoietin stimulating agent (ESA) or a HIF-PHI within 12 weeks of informed consent
11. History of malignant hypertension or current uncontrolled hypertension (average systolic blood pressure ≥ 160 mmHg and/or average diastolic blood pressure ≥ 100 mmHg based on 3 readings). Blood pressure should be measured after 5 minutes of unattended rest, with 2 repeated readings 1 to 2 minutes apart
12. History of diabetic retinopathy
13. History or diagnosis of any of the following:

    1. Anemia due to pernicious anemia, thalassemia, sickle cell anemia, sickle trait, or myelodysplastic syndromes
    2. Bone-marrow hypoplasia or pure red cell aplasia
    3. Androgen deprivation therapy within the previous 12 months or radiation treatment for prostate cancer
    4. Myocardial infarction, acute coronary syndrome, stroke, transient ischemic attack, or prothrombotic arrhythmia or condition (e.g., untreated/uncontrolled atrial fibrillation) within 6 months before informed consent or during the Screening Period
    5. Active malignancy and/or receiving anti cancer treatment within 12 weeks of informed consent (squamous cell or basal cell carcinoma of the skin are excluded from this criterion). Subjects who have planned initiation of cancer therapies during the study period (such as, but not limited to, chemotherapy, radiotherapy) are excluded.
14. Planned intravenous (IV) iron therapy scheduled to start after informed consent and to continue during the expected time of participation in the study
15. Presence of acute kidney injury (AKI) based upon the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines:

    1. Increase in serum creatinine by ≥ 0.3 mg/dL (≥ 26.5 µmol/L) within 48 hours, or
    2. Increase in serum creatinine to ≥ 1.5 times the value at baseline, which is known or presumed to have occurred within the previous 7 days
16. Chronic bleeding condition such as active gastrointestinal (GI) bleeding
17. Inability or unwillingness to adhere to protocol specified visits, procedures, and contraception requirements
18. Receipt of an investigational drug or device within 30 days before informed consent
19. Previously screened for or enrolled in the BGE-117-203 study
20. Known allergy to or intolerance of BGE-117, or other components of the IP (BGE-117 or matching placebo)
21. Known allergy to ferrous sulfate preparations

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Time to 2.0 g/dL Increase in Hemoglobin Level | Up to Day 85
  The time to a 2.0 g/dL increase in hemoglobin level over the postoperative baseline hemoglobin level. The primary comparison is the high-dose group compared to placebo.
  Note: Baseline hemoglobin level is the postoperative hemoglobin level most recently obtained before the start of investigational product administration.

SECONDARY OUTCOMES:
Hemoglobin Level from Baseline | Day 8, 15, 22, 29, 36, 43, 57, and 85
  Change in hemoglobin level from baseline.
Hemoglobin Level from Nadir Hemoglobin | Day 8, 15, 22, 29, 36, 43, 57, and 85
  Change in hemoglobin level from nadir hemoglobin.
Time to 1.0 g/dL Increase in Hemoglobin Level | Up to Day 85
  The time to a 1.0 g/dL increase in hemoglobin level over the postoperative baseline hemoglobin level.
  Note: Baseline hemoglobin level is the postoperative hemoglobin level most recently obtained before the start of investigational product administration.
Time to 3.0 g/dL Increase in Hemoglobin Level | Up to Day 85
  The time to a 3.0 g/dL increase in hemoglobin level over the postoperative baseline hemoglobin level.
  Note: Baseline hemoglobin level is the postoperative hemoglobin level most recently obtained before the start of investigational product administration.
Hemoglobin Level Return to Baseline for Elective Hip Replacement | Day 8, 15, 22, 29, 36, 43, 57, and 85
  Proportion of elective hip replacement subjects who return to preoperative baseline hemoglobin level.
1.0 g/dL Improvement in Hemoglobin Level | Day 8, 15, 22, 29, 36, 43, 57, and 85
  Proportion of subjects with a 1.0 g/dL improvement in hemoglobin level from the postoperative baseline hemoglobin value
2.0 g/dL Improvement in Hemoglobin Level | Day 8, 15, 22, 29, 36, 43, 57, and 85
  Proportion of subjects with a 2.0 g/dL improvement in hemoglobin level from the postoperative baseline hemoglobin value
3.0 g/dL Improvement in Hemoglobin Level | Day 8, 15, 22, 29, 36, 43, 57, and 85
  Proportion of subjects with a 3.0 g/dL improvement in hemoglobin level from the postoperative baseline hemoglobin value
All-Cause Mortality | First Dose to Day 85 and Follow-up (Up to Day 183)
  The rate of all-cause mortality.
Hospital Readmission - Any Cause | First Dose to Day 85 and Follow-up (Up to Day 183)
  The rate of hospital readmissions for any cause.
Hospital Readmission - Surgery-Related | First Dose to Day 85 and Follow-up (Up to Day 183)
  The rate of hospital readmissions for causes related to surgery.
Surgical Complications | First Dose to Day 85 and Follow-up (Up to Day 183)
  The rate of surgical complications (e.g., dislocation, nonunion, infection, chronic pain, posttraumatic arthritic changes, avascular necrosis).
Surgical Complications by Clavien-Dindo Classification | First Dose to Day 85 and Follow-up (Up to Day 183)
  The rate of surgical complications as defined by the Clavien-Dindo Classification of ≥ Grade II Defined as follows:
  Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Grade III-IIIB: Requiring surgical, endoscopic or radiological intervention. Intervention not under general anesthesia. Intervention under general anesthesia.
  Grade IV-IVb: Life-threatening complication (including CNS complications) requiring IC/ICU-management. Single organ dysfunction (including dialysis). Multiorgan dysfunction.
  Grade V: Death of a patient.
Change in Ambulation Status | First Dose to Day 85 and Follow-up (Up to Day 183)
  The time to change in ambulation status (e.g., from ambulation with human assistance to ambulation with assistive device, or to independent ambulation).
Days Alive and At Home (DAH) | Day 30
  Number of days that the subject has been at home. Home is defined as the subject's place of residence before surgery.
Days Alive and At Home (DAH) | Day 60
  Number of days that the subject has been at home. Home is defined as the subject's place of residence before surgery.
Analysis of Pharmacokinetic Parameters to Develop a Population Pharmacokinetic Model for BGE-117 (AUC(0-24)/Dose) | Day 1, 43, and 85
  Single blood samples for pharmacokinetic analysis will be collected just prior to first dose and on Days 43 and 85. Time of last dose and time of blood draw will be collected and these data will be used to attempt to develop a population pharmacokinetic model of BGE-117. If possible, AUC(0-24)/dose will be determined. Age, gender and renal function will be explored as covariates.
Analysis of Pharmacokinetic Parameters to Develop a Population Pharmacokinetic Model for BGE-117 (Clearance) | Day 1, 43, and 85
  Single blood samples for pharmacokinetic analysis will be collected just prior to first dose and on Days 43 and 85. Time of last dose and time of blood draw will be collected and these data will be used to attempt to develop a population pharmacokinetic model of BGE-117. If possible, clearance will be determined. Age, gender and renal function will be explored as covariates.
Analysis of Pharmacokinetic Parameters to Develop a Population Pharmacokinetic Model for BGE-117 (Volume of Distribution) | Day 1, 43, and 85
  Single blood samples for pharmacokinetic analysis will be collected just prior to first dose and on Days 43 and 85. Time of last dose and time of blood draw will be collected and these data will be used to attempt to develop a population pharmacokinetic model of BGE-117. If possible, volume of distribution will be determined. Age, gender and renal function will be explored as covariates.
Analysis of Pharmacokinetic Parameters to Develop a Population Pharmacokinetic Model for BGE-117 (Half-Life) | Day 1, 43, and 85
  Single blood samples for pharmacokinetic analysis will be collected just prior to first dose and on Days 43 and 85. Time of last dose and time of blood draw will be collected and these data will be used to attempt to develop a population pharmacokinetic model of BGE-117. If possible, half-life will be determined. Age, gender and renal function will be explored as covariates.
Subjects Requiring a Dose Decrease | Up to Day 85
  The proportion of subjects requiring a decrease in the investigational product dose. Dose decreases are allowed for safety, tolerability, and to maintain an approximate rate of hemoglobin increase of ≤ 1.5 g/dL every 2 weeks, and a maximum hemoglobin level of 12.0 g/dL.
Mean Dose at End of Study | Day 85
  The mean dose at the end of the treatment period including any dose decreases and/or termination of dose.
Disposition after Hospital Discharge | Up to Day 85
  The location where the subject is discharged following discharge from the hospital (e.g., home, rehabilitation center, nursing-care facility, etc.)
Hemoglobin Response as a Function of Iron Status and Hepcidin | Up to Day 85
  The rate of hemoglobin level increase as a function of subject baseline iron status and hepcidin.
Hemoglobin Response as a Function of Clinical Outcome Assessment | Up to Day 85
  The rate of hemoglobin level increase as a function of the results from defined clinical outcome assessments (QoR-15 questionnaire, VAS-pain related to the surgical site, WHODAS, EQ-5D-5L, 6MWT, TUG test)
Quality of Recovery-15 (QoR-15) Questionnaire | Day 8, 15, 22, and 29
  Change in QoR-15 Questionnaire compared to baseline. The QoR-15 questionnaire is a 15 item questionnaire used to evaluate postoperative quality of recovery in the areas of pain, physical comfort, physical independence, psychological support and emotional state. Each question is scored from 0 (very poor recovery) to 10 (excellent recovery). A higher score is considered a better outcome.
Visual Analog Scale for Pain (VAS-Pain) | Up to Day 15
  Change in VAS-Pain compared to baseline. The VAS-Pain is used to assess the subject's pain at the surgical site at that moment in time. The scale is from 0 (no pain) to 10 (extreme pain). A lower score is considered a better outcome.
World Health Organization Disability Assessment Schedule (WHODAS) Questionnaire | Day 29, 57, and 85
  Change in WHODAS Questionnaire compared to baseline. The WHODAS is a general health status questionnaire designed to produce standardized disability levels by elucidating the subject's perception of health on several domains, including cognition, mobility, self-care, getting along, life activities (household and work), and participation. The questionnaire contains 36 questions that ask the subject to recall difficulty in performing activities he/she felt during the previous 30 days. The scale is from 1 (none) to 5 (extreme or cannot do). A lower score is considered a better outcome.
European Quality of Life Five Day (EQ-5D-5L) Questionnaire | Day 15, 43, and 85
  Change in EQ-5D-5L Questionnaire compared to baseline. The EQ-5D-5L questionnaire is a 5 question tool used to assess treatment effects by measuring the gains (or losses) in subject-reported health status. The questionnaire assesses five dimensions: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each item is scored on a scale from 1 (no problems) to 5 (extreme or cannot perform). A lower score is considered a better outcome.
6-minute Walk Test (6MWT) Distance | Day 15, 43, and 85
  Change in 6MWT Distance compared to baseline. Increased distance is considered a better outcome.
Timed Up and Go (TUG) Test | Day 15, 43, and 85
  Change in TUG test time compared to baseline. The TUG test is used to assess mobility and consists of the subject standing up from a chair, walking 3 meters away, turning, walking back 3 meters, and sitting down again. A shorter time is considered a better outcome.
Safety Analyses (Treatment-Emergent Adverse Events) - Incidence | First Dose to Day 85 and Follow-up (Up to Day 183)
  Safety analyses will be performed based on the corresponding safety set. The incidence of treatment-emergent AEs (TEAEs) will be calculated overall by system organ class, preferred term, and treatment group for each cohort and treatment group. The number and percentage of subjects with TEAEs will be further summarized by severity and relationship to the investigational product and dose level.
Safety Analyses (Treatment-Emergent Adverse Events) - Number of Events | First Dose to Day 85 and Follow-up (Up to Day 183)
  Safety analyses will be performed based on the corresponding safety set. The number of events of treatment-emergent AEs (TEAEs) will be calculated overall by system organ class, preferred term, and treatment group for each cohort and treatment group. The number of subjects with TEAEs will be further summarized by severity and relationship to the investigational product and dose level.
Safety Analyses (Treatment-Emergent Adverse Events) - Percentage | First Dose to Day 85 and Follow-up (Up to Day 183)
  Safety analyses will be performed based on the corresponding safety set. The percentage of treatment-emergent AEs (TEAEs) will be calculated overall by system organ class, preferred term, and treatment group for each cohort and treatment group. The percentage of subjects with TEAEs will be further summarized by severity and relationship to the investigational product and dose level.
Safety Analyses (Adverse Events) - Individual Summary | First Dose to Day 85 and Follow-up (Up to Day 183)
  Adverse events related to investigational product, AEs leading to withdrawal, SAEs, and deaths will be summarized/listed as part of the overall analysis of safety.
Safety Analyses (Quantitative Safety Data) - Clinical Laboratory Tests | First Dose to Day 85 and Follow-up (Up to Day 183)
  Clinical laboratory tests (complete blood count, HemoCue, serum clinical chemistries, coagulation, serum erythropoietin levels, hemoglobin electrophoresis, inflammation panel, iron panel, folate and vitamin B12, lipid panel, thyroid, and urinalysis) findings will be summarized by treatment group and visit. Descriptive statistics will be calculated for quantitative safety data as well as for the difference from baseline, if applicable. Frequency counts will be compiled for the classification of qualitative safety data. The baseline for safety data will be defined as the last value prior to the first dose of investigational product. Potentially clinically important findings will also be summarized or listed.
Safety Analyses (Quantitative Safety Data) - Vital Signs | First Dose to Day 85 and Follow-up (Up to Day 183)
  Vital signs (systolic and diastolic blood pressure and pulse rate) findings will be summarized by treatment group and visit. Descriptive statistics will be calculated for quantitative safety data as well as for the difference from baseline, if applicable. Frequency counts will be compiled for the classification of qualitative safety data. The baseline for safety data will be defined as the last value prior to the first dose of investigational product. Potentially clinically important findings will also be summarized or listed.
Safety Analyses (Quantitative Safety Data) - Wells Score for DVT | First Dose to Day 85 and Follow-up (Up to Day 183)
  The Well's Criteria will be used to evaluate for the presence of deep vein thrombosis (DVT) and summarized by treatment group and visit. Descriptive statistics will be calculated for quantitative safety data as well as for the difference from baseline, if applicable. Frequency counts will be compiled for the classification of qualitative safety data. The baseline for safety data will be defined as the last value prior to the first dose of investigational product. Potentially clinically important findings will also be summarized or listed.
Safety Analyses (Quantitative Safety Data) - Electrocardiogram (ECG) | First Dose to Day 85 and Follow-up (Up to Day 183)
  Electrocardiogram (ECG) will be performed with heart rate, PR, QRS, and QT (pre-corrected) intervals will be measured and QTcF will be calculated. ECG findings will be summarized by treatment group and visit. Descriptive statistics will be calculated for quantitative safety data as well as for the difference from baseline, if applicable. Frequency counts will be compiled for the classification of qualitative safety data. The baseline for safety data will be defined as the last value prior to the first dose of investigational product. Potentially clinically important findings will also be summarized or listed.

OTHER OUTCOMES:
Days Alive and At Home (DAH) | Day 90
  Number of days that the subject has been at home. Home is defined as the subject's place of residence before surgery.
Days Alive and At Home (DAH) | Day 120
  Number of days that the subject has been at home. Home is defined as the subject's place of residence before surgery.
Days Alive and At Home (DAH) | Day 183
  Number of days that the subject has been at home. Home is defined as the subject's place of residence before surgery.
Hemoglobin Level from Baseline | Day 99, 127, 155 and 183
  Change in hemoglobin level from baseline.
Hemoglobin Level from Nadir Hemoglobin | Day 99, 127, 155 and 183
  Change in hemoglobin level from nadir hemoglobin.
Subjects Who are Non-anemic per WHO Criteria | Day 99, 127, 155 and 183
  The proportion of subjects who are non-anemic by WHO criteria (Hemoglobin of ≥12 g/dL for women, ≥13 g/dL for men).
Hemoglobin Level Return to Baseline for Elective Hip Replacement | Day 99, 127, 155, and 183
  Proportion of elective hip replacement subjects who return to preoperative baseline hemoglobin level.
Subjects with 2.0 g/dL Increase in Hemoglobin Level | Day 99, 127, 155, and 183
  Proportion of subjects with a ≥2.0 g/dL increase in hemoglobin level.
Visual Analog Scale for Pain (VAS-Pain) | Day 183
  Change in VAS-Pain compared to baseline. The VAS-Pain is used to assess the subject's pain at the surgical site at that moment in time. The scale is from 0 (no pain) to 10 (extreme pain). A lower score is considered a better outcome.
World Health Organization Disability Assessment Schedule (WHODAS) Questionnaire | Day 183
  Change in WHODAS Questionnaire compared to baseline. The WHODAS is a general health status questionnaire designed to produce standardized disability levels by elucidating the subject's perception of health on several domains, including cognition, mobility, self-care, getting along, life activities (household and work), and participation. The questionnaire contains 36 questions that ask the subject to recall difficulty in performing activities he/she felt during the previous 30 days. The scale is from 1 (none) to 5 (extreme or cannot do). A lower score is considered a better outcome.
European Quality of Life Five Day (EQ-5D-5L) Questionnaire | Day 183
  Change in EQ-5D-5L Questionnaire compared to baseline. The EQ-5D-5L questionnaire is a 5 question tool used to assess treatment effects by measuring the gains (or losses) in subject-reported health status. The questionnaire assesses five dimensions: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each item is scored on a scale from 1 (no problems) to 5 (extreme or cannot perform). A lower score is considered a better outcome.
Occurrence of Wound Dehiscence | Up to Day 85
  The rate of occurrence for wound dehiscence from the index surgery to the end of investigational product administration.
Occurrence of Surgical Site Infections (SSIs) | Up to Day 85
  The rate of occurrence for SSIs from the index surgery to the end of investigational product administration.
Bone Healing at Surgical Site | Day 183
  The level of bone healing at the surgical site compared to baseline by radiographic evidence.
Scar Formation/Quality | Up to Day 85
  The scar formation/quality assessed at the end of IP administration. The assessment is done by Vancouver scar scale and the Patient and Observer Scar Assessment Scale (POSAS). The Vancouver scar scale assesses scar vascularity, pigmentation, pliability and height. A lower score is considered a better outcome. The POSAS assesses the scar by pain, itch, thickness, color, stiffness and irregularity. A lower score is considered a better outcome.
Activity Level and Sleep Quality | Up to Day 183
  The subjects' activity level and sleep quality are measured by a wearable activity monitor. These data may be algorithmically transformed into a number of exploratory endpoints, including, but not limited to, time spent in light, moderate, or vigorous activity, or in combinations thereof such as moderate to vigorous activity; time spent sedentary or in locomotion; estimated calories expended; total motion in each spatial axis or in all spatial axes; number of steps taken; time spent sleeping; the number of or length of awakenings during a sleep period; and the proportion of each overall sleep period (including temporary awakenings) spent in sleep or time in each overall sleep period (including temporary awakenings) spent in sleep.
Iron Status Effect | Up to Day 183
  Evaluate the effect of iron status at baseline on the response to investigational product administration and change in iron parameters throughout the study.
Inflammation Markers Effect | Up to Day 85
  Evaluate the effect of Markers of Inflammation (hepcidin, C-Reactive Protein [CRP], interleukin [IL-1, IL-6], and tumor necrosis factor alpha [TNF- α]) at baseline on the response to investigational product administration and change in inflammatory markers during investigational product administration.
Postoperative Iron Stores Effect | Up to Day 183
  Evaluate the effect of status of postoperative iron stores on the response to investigational product administration throughout the study.
Patient-Reported Outcomes and Anemia Response Correlation | Up to Day 183
  Evaluate correlations of various functional patient-reported outcomes (e.g., WHODAS, EQ-5D-5L, etc.) to the therapeutic response (e.g., hemoglobin increase) at various timepoints.

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Research, Gosford, New South Wales, Australia